CLINICAL TRIAL: NCT00605644
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Oral MOA-728 for the Treatment of Opioid-Induced Bowel Dysfunction in Subjects With Chronic Nonmalignant Pain
Brief Title: Study Evaluating MOA-728 Oral for the Treatment of OIBD in Subjects With Chronic Non-Malignant Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3200A3-2202
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 150 mg (Experimental): MOA-728
  Interventions: Drug: MOA-728
- 300 mg (Experimental): MOA-728
  Interventions: Drug: MOA-728
- 450 mg (Experimental): MOA-728
  Interventions: Drug: MOA-728
- 600 mg (Experimental): MOA-728
  Interventions: Drug: MOA-728

INTERVENTIONS:
Drug: MOA-728 — Oral Capsules
  Arms: 150 mg; 300 mg; 450 mg; 600 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and dose-response relationship of N-methylnaltrexone bromide (MOA-728) by observing spontaneous bowel movements in subjects administered MOA-728 who have chronic pain that is not due to cancer, and who have opioid-induced bowel dysfunction (OIBD).

ELIGIBILITY:
Inclusion Criteria:

* Adult Outpatients with opioid-induced bowel dysfunction and chronic pain, which is not due to malignant cancer.
* Taking oral, transdermal, intravenous, or subcutaneous opioids.
* Willingness to discontinue all pre-study laxative therapy and use only study permitted rescue laxatives.

Exclusion Criteria:

* History of chronic constipation before the initiation of opioid therapy.
* Other GI disorders known to affect bowel transit.
* Women who are pregnant, breast feeding, or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg
Started | 29 | 19 | 20 | 30 | 30
Completed | 28 | 18 | 18 | 25 | 22
Not Completed | 1 | 1 | 2 | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg | Total
Number analyzed (Participants) | 29 | 19 | 20 | 30 | 30 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.24 (10.45) | 54.68 (9.49) | 51.25 (12.72) | 50.17 (10.46) | 49.13 (8.59) | 51.69 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 9 | 10 | 18 | 22 | 77
  Male | 11 | 10 | 10 | 12 | 8 | 51

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Witn Spontaneous Bowel Movements Within 3 Hours of Treatment
Time Frame: 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg
Number analyzed (Participants) | 29 | 19 | 20 | 30 | 30
Participants | 2 | 3 | 2 | 5 | 6

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Placebo | 150 mg | 300 mg | 450 mg | 600 mg
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/19 | 0/20 | 1/30 | 2/30
Other Adverse Events (participants affected / at risk) | 4/29 | 3/19 | 9/20 | 12/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | 150 mg (N=19) | 300 mg (N=20) | 450 mg (N=30) | 600 mg (N=30)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | 150 mg (N=19) | 300 mg (N=20) | 450 mg (N=30) | 600 mg (N=30)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Haemorrhoid (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1
Pyrexia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Band neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.